CLINICAL TRIAL: NCT06298630
Title: Long-term Follow-up Study of BRL-101 in the Treatment of Transfusion-dependent β-thalassemia
Brief Title: Long-term Follow-up Study of BRL-101 for TDT
Status: Not yet recruiting | Type: Observational
Sponsor: Bioray Laboratories (Industry)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Xiangya Hospital of Central South University (Other); Chinese Academy of Medical Sciences (Other); Nanfang Hospital, Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other); Shenzhen Children 's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-LTF-BRL-101
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: Thalassemia, Beta
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BRL-101: All patients who have received BRL-101
  Interventions: Other: Assessments

INTERVENTIONS:
Other: Assessments — Safety and efficacy assessments

SUMMARY:
Observe long-term safety risk and long-term efficacy after intravenous infusion of BRL-101 in TDT subjects.

DETAILED DESCRIPTION:
Observe long-term delayed safety risks such as emerging neoplasms, emerging haematological disorders, and long-term efficacy after intravenous infusion of BRL-101 in TDT subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent for this study by subjects, or as applicable, subject's parent(s)/legal guardian(s)
2. Treated with BRL-101 for therapy of transfusion-dependent β-thalassemia.

Exclusion Criteria:

- There are no exclusion criteria for this study

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with transfusion-dependent β-thalassemia who have been treated with BRL-101.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-08 (Estimated); Primary Completion 2038-08-20 (Estimated); Study Completion 2038-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of hematologic malignancies | Up to 15 years post-drug product infusion
  Such as new lymphoma, leukemia, MDS, etc.
Frequency, grade, and relationship of SAEs | Within 2 years to 5years after BRL-101 Infusion
  Frequency, grade, and relationship to BRL-101 of SAEs following BRL-101 reinfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochen Wang, Study Chair — Bioray Laboratories
Locations (7):
- China (7):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen Children 's Hospital, Shenzhen, Guangdong
  - No. 923 Hospital of Joint Support Force of Chinese People 's Liberation Army Hospital, Nanning, Guangxi
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Tianjin Institute of Hematology, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of GUANGXI MEDICAL UNIVERSITY, Guangxi

IPD SHARING:
Plan to Share IPD: Undecided